CLINICAL TRIAL: NCT04226833
Title: An Open-Label, One Treatment, Four Group, Parallel Group Study to Investigate the Effect of Impaired Hepatic Function on the Pharmacokinetics of Entrectinib in Volunteers With Different Levels of Hepatic Function
Brief Title: A Study to Investigate the Effect of Impaired Hepatic Function on the Pharmacokinetics of Entrectinib in Volunteers With Different Levels of Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP41174; 2019-003065-17 (EudraCT Number)
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Insufficiency
Keywords: Hepatic Impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — entrectinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild (Experimental): Participants with mild hepatic impairment will receive 1x100 milligram (mg) F06 (entrectinib) capsule administered orally with approximately 240 milliliter (mL) water within 30 minutes after consumption of a standardized meal.
  Interventions: Drug: entrectinib
- Moderate (Experimental): Participants with moderate hepatic impairment will receive 1x100 mg F06 (entrectinib) capsule administered orally with approximately 240 mL water within 30 minutes after consumption of a standardized meal.
  Interventions: Drug: entrectinib
- Severe (Experimental): Participants with severe hepatic impairment will receive 1x100 mg F06 (entrectinib) capsule administered orally with approximately 240 mL water within 30 minutes after consumption of a standardized meal.
  Interventions: Drug: entrectinib
- Normal (Experimental): Participants with normal hepatic function will receive 1x100 mg F06 (entrectinib) capsule administered orally with approximately 240 mL water within 30 minutes after consumption of a standardized meal.
  Interventions: Drug: entrectinib

INTERVENTIONS:
Drug: entrectinib — 1x100 milligram (mg) capsule given with approximately 240 milliliter (mL) of water within 30 minutes of consumption of a standardized meal
  Other Names: F06 formulation; Rozlytrek

SUMMARY:
This is a non-randomized, open-label, one treatment, four group, parallel group study to investigate the effect of impaired hepatic function on the pharmacokinetics of entrectinib in participants with different levels of hepatic function. Participants with mild, moderate or severe hepatic impairment ('Mild', 'Moderate' and 'Severe' groups), and control participants with normal hepatic function ('Normal' group) will each receive a single 100 mg dose of entrectinib after consumption of a standardized meal.

DETAILED DESCRIPTION:
Participants with reduced hepatic function will be assigned to a functional category based on assessments at the Screening visit. Each individual will be categorized according to the Child Pugh system for classifying hepatic impairment and also according to the National Cancer Institute organ dysfunction working group (NCI-ODWG) system. Recruitment will be staggered to allow review of pharmacokinetic and safety data from at least three participants in each of the Mild and Moderate groups before participants are enrolled into the Severe group. Recruitment of the Severe group will only proceed if there is agreement between the Sponsor and the Investigator that data from this group are necessary to fulfill the objectives of the study and that dosing is not anticipated to present an unacceptable risk to those individuals. The control group of participants with normal hepatic function will be enrolled after the full complement of participants with hepatic dysfunction has been dosed.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* A body mass index (BMI) between 18.0 and 38.0 kg/m2, and weighing at least 50 kg
* Agreement to comply with measures to prevent pregnancy and restrictions on sperm donation.

Participants with normal hepatic function:

* Normal hepatic function and no history of clinically significant hepatic dysfunction.
* Healthy for age-group in the opinion of the Investigator.

Participants with hepatic impairment:

* Mild, moderate or severe hepatic dysfunction (i.e. Child-Pugh A, B or C, NCIODWG Mild, Moderate or Severe) arising from cirrhosis of the liver as the result of parenchymal liver disease.
* Stable hepatic function.

Exclusion Criteria:

* Transjugular intrahepatic portosystemic shunt or other porta-caval shunt.
* A history of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers.
* Recent history or signs of severe hepatic encephalopathy (e.g., a portal systemic encephalopathy score >2).
* Advanced ascites or ascites which require emptying and albumin supplementation.
* Hepatocellular carcinoma, acute liver disease or serum ALT or AST not consistent with stable disease.
* Recipient of a liver transplant.
* Uncontrolled hypertension.
* Clinically significant impairment of renal function.
* A history of gastrointestinal surgery or other gastrointestinal disorder that might affect absorption of medicines from the gastrointestinal tract.
* Clinically significant change in health status, or any major illness, or clinically significant acute infection or febrile illness.
* Women who are pregnant or lactating.
* Presence of any abnormal ECG finding, which is clinically significant.
* Use of moderate or potent inhibitors or inducers of cytochrome P450 3A4 enzyme.
* Participation in any other clinical study involving administration of an investigational medicinal product or use of an unapproved device.
* A positive test result for human immunodeficiency virus (HIV).
* Known history of clinically significant hypersensitivity, or severe allergic reaction, to entrectinib or related compounds or other excipients in the entrectinib formulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Pharmaceutical Research Associates CZ, s.r.o., Prague, Czechia
- CRU Hungary Kft, Miskolc, Hungary
- Summit Clinical Research s.r.o.; Oddelenie internej mediciny a klinickej farmakologie, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Ozbey AC, Meneses-Lorente G, Simmons B, McCallum S, Annaert P, Parrott N, Umehara K. Clinical Exploration and Physiologically Based Modelling of the Impact of Hepatic Impairment on Entrectinib Pharmacokinetics. Clin Pharmacokinet. 2025 Mar;64(3):437-451. doi: 10.1007/s40262-024-01468-y. Epub 2025 Feb 11. PMID 39934586

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with reduced hepatic function were assigned to a functional category based on assessments at the Screening visit.
Period: Overall Study
Arm/Group | Mild | Moderate | Severe | Normal
Started | 7 | 12 | 11 | 8
Completed | 7 | 12 | 10 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild | Moderate | Severe | Normal | Total
Number analyzed (Participants) | 7 | 12 | 11 | 8 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (8.86) | 58.0 (9.49) | 57.3 (10.08) | 54.3 (11.99) | 57.3 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 3 | 9
  Male | 5 | 9 | 10 | 5 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 12 | 11 | 8 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Entrectinib
Description: Maximum observed plasma concentration. Observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
nmol/L | 296.140 (40.6) | 213.570 (36.7) | 183.680 (34.3) | 235.990 (46.1)

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE=adverse event TEAE=treatment-emergent adverse event
Time Frame: 4 weeks
Measure: Number; unit: Participants
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
Participants
  Total Subjects With at Least 1 AE | 0 | 1 | 2 | 2
  Subjects With at Least 1 TEAE | 0 | 1 | 2 | 2
  Total Subjects with at Least 1 Serious TEAE | 0 | 0 | 1 | 0

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUCinf) of Entrectinib
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h*nmol/L | 5525.6 (47.0) | 5401.9 (49.1) | 6329.0 (58.5) | 3512.7 (50.8)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUClast) of Entrectinib
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h*nmol/L | 5263.9 (48.4) | 4952.3 (49.0) | 5747.9 (53.6) | 3283.2 (51.5)

5. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Entrectinib
Description: First observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units
Time Frame: From Day 1 to Day 7
Measure: Median (Full Range); unit: h
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h | 4.000 [2.05 to 4.83] | 5.000 [2.95 to 8.05] | 3.000 [1.00 to 5.97] | 2.950 [1.00 to 4.88]

6. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Entrectinib
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h | 30.75 (18.7) | 30.43 (36.5) | 43.92 (30.2) | 21.34 (36.8)

7. Primary Outcome: Apparent Terminal Elimination Rate Constant (Lz) of Entrectinib
Time Frame: From Day 1 to Day 7
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
1/h | 0.0229 (0.00430) | 0.0241 (0.00858) | 0.0165 (0.00544) | 0.0345 (0.01359)

8. Primary Outcome: Apparent Oral Clearance (CL/F) of Entrectinib
Description: Obtained by dividing the total dose of parent drug by its corresponding AUCinf
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/(h*nmol/L)
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
mg/(h*nmol/L) | 0.0200 (47.0) | 0.0200 (49.1) | 43.92 (30.2) | 0.0300 (50.8)

9. Primary Outcome: The Apparent Volume of Distribution (Vz/F) of Entrectinib
Description: Obtained by dividing Dose by the product of AUCinf and λz
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/(nmol/L)
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
mg/(nmol/L) | 0.8000 (47.7) | 0.8100 (37.6) | 1.0000 (35.2) | 0.8800 (43.8)

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of M5
Description: as for outcome 1
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
nmol/L | 41.310 (71.0) | 26.390 (68.6) | 17.710 (58.3) | 60.330 (41.7)

11. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUCinf) of M5
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h*nmol/L | 2432.1 (17.2) | 2024.3 (58.8) | NA (NA) — Below the level of detection | 2229.9 (40.3)

12. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUClast) of M5
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h*nmol/L | 1255.2 (67.8) | 1297.3 (52.4) | 1202.8 (62.9) | 1715.6 (48.7)

13. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of M5
Description: as for outcome 5
Time Frame: From Day 1 to Day 7
Measure: Median (Full Range); unit: h
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h | 5.000 [4.83 to 8.00] | 5.955 [3.00 to 35.50] | 4.920 [2.83 to 71.80] | 4.985 [2.98 to 7.97]

14. Primary Outcome: Apparent Terminal Elimination Rate Constant (Lz) of M5
Time Frame: From Day 1 to Day 7
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
1/h | 0.02000 (2.5) | 0.0200 (30.4) | NA (NA) — Below the level of detection | 0.0200 (22.8)

15. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of M5
Time Frame: From Day 1 to Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 7 | 12 | 11 | 8
h | 43.60 (2.5) | 39.50 (30.4) | NA (NA) — Below the level of detection | 38.33 (22.8)

ADVERSE EVENTS:
Time Frame: Baseline up to 4 Weeks
Groups:
- Entrectinib - Normal; Entrectinib Mild; Entrectinib Moderate; Entrectinib Severe: Participants received 1x100 milligram (mg) F06 (entrectinib) capsule administered orally with approximately 240 milliliter (mL) water within 30 minutes after consumption of a standardized meal.
Arm/Group | Entrectinib - Normal | Entrectinib Mild | Entrectinib Moderate | Entrectinib Severe
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/12 | 1/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 2/8 | 0/7 | 1/12 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entrectinib - Normal (N=8) | Entrectinib Mild (N=7) | Entrectinib Moderate (N=12) | Entrectinib Severe (N=11)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entrectinib - Normal (N=8) | Entrectinib Mild (N=7) | Entrectinib Moderate (N=12) | Entrectinib Severe (N=11)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT04226833/Prot_SAP_000.pdf